CLINICAL TRIAL: NCT01868386
Title: Hypofractionated Post-prostatectomy Radiotherapy for Prostate Cancer to Reduce Toxicity and Improve Patient Convenience: A Phase I/II Trial
Brief Title: Shorter Duration Radiotherapy to Treat Prostate Cancer After Removal of the Prostate
Acronym: HypoFX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Timothy Showalter, MD (Other)
Responsible Party: Sponsor-Investigator, Timothy Showalter, MD, Professor, Radiation Oncology, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16604
Record Dates: First submitted 2013-05-14; First posted 2013-06-04 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Radiotherapy, hypofractionated; Salvage therapy; Radiotherapy, adjuvant
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 1 (Experimental): Hypofractionated therapy, 26 treatments at 2.5 Gy
  Interventions: Radiation: Hypofractionated therapy
- Dose Level 2 (Experimental): Hypofractionated therapy, 20 treatments at 2.83Gy
  Interventions: Radiation: Hypofractionated therapy
- Dose Level 3 (Experimental): Hypofractionated therapy,15 treatments at 3.36 Gy
  Interventions: Radiation: Hypofractionated therapy
- Dose Level 4 (Experimental): Hypofractionated therapy, 10 treatments at 4.26 Gy
  Interventions: Radiation: Hypofractionated therapy

INTERVENTIONS:
Radiation: Hypofractionated therapy — Shorter courses of increasing doses of radiation therapy will be assessed in each subsequent arm

SUMMARY:
Radiation therapy is one of the standard treatments for men with prostate cancer who have detectable levels of prostate specific antigen (PSA, a prostate cancer specific marker) after surgery. When radiation therapy is given to patients who have an increase in PSA after surgery, it is called "salvage radiation therapy". Currently the standard radiation therapy course length for this type of cancer is around 7 ½ -8 weeks. Sometimes, radiation therapy after prostate removal causes unpleasant side effects. A shorter course of radiation therapy, known as a "hypofractionated" course, gives fewer but higher doses of radiation than standard radiation.

The purpose of this study is to test the safety of a shorter course of radiation therapy at progressively lower dose levels and shorter lengths of treatment (hypofractionated) with patients who have had their prostate removed. The study will assess whether the hypofractionated course works better without causing additional side effects to the remaining cancer cells in the prostate bed.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the shortest dose-fractionation schedule (Dose Schedule) with acceptable grade ¡Ã 3 GU/GI toxicity rate for salvage HypoFx RT to maintain a constant, high BED for prostate cancer response while reducing the BED for late GU and GI toxicity

To assess health-related quality of life (HRQOL) of the recommended Dose Schedule of salvage HypoFx RT by demonstrating no significant change in 1-year disease specific QoL, as compared to baseline

Secondary Objectives:

To evaluate and characterize the acute and late genitourinary (GU) and gastrointestinal (GI) adverse effects associated with postoperative, hypofractionated radiation therapy.

To evaluate biochemical failure rate, defined separately as nadir plus 2 ng/mL and as three consecutive rises in PSA, at 2 years after hypofractionated, post-prostatectomy radiation therapy.

To evaluate health utilities at 1 year after HypoFx salvage RT, as measured by the EQ-5D instrument.

To evaluate changes in sexual domain of EPIC quality of life instrument at 1 year after HypoFx salvage RT.

To evaluate the treatment burden for patients undergoing salvage HypoFx RT, in order to examine whether HypoFx RT results in less burdensome treatment for patients, as measured by patient-reported direct and indirect (i.e., transportation) health care costs and lost productivity due to treatment, as evaluated by the Work Productivity and Activity Impairment Questionnaire¢-General Health (WPAI-GH).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of prostate adenocarcinoma and
* have had a prostatectomy
* have detectable PSA
* 18 years of age or older

Exclusion Criteria:

* are receiving chemotherapy or other agents intended for cancer treatment
* history of rectal surgery or lower gastrointestinal bleed
* history of bleeding diathesis or abnormal sensitivity to ionizing radiation
* had prior pelvic irradiation or are scheduled to receive pelvic nodal irradiation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | over a period of 2 years
  Incidence of GU (genitourinary) and GI (gastrointestinal) toxicities of CTCAE (Common Terminology Criteria for Adverse Events) grade 3 or greater
Quality of life measure | over a period of 2 years
  To compare quality of life post-procedure from baseline

SECONDARY OUTCOMES:
Biochemical failure rate | over a period of 2 years
  A biochemical failure is defined as an increase in prostate serum antigen concentration to nadir plus 2ng/mL or 3 consecutive increases in PSA

OTHER OUTCOMES:
Acute and late GU and GI toxicity | over a period of two years
Health Utilities | 1 year after radiation treatment
EPIC Prostate Cancer-Specific QOL instrument | over a period of two years
  looking at changes in sexual and hormonal domains
Ancillary financial burden | over a period of two years
  estimating out-of-pocket costs and lost wages for patients during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Showalter, MD, Principal Investigator — University of Virginia School of Medicine
Locations (3):
- United States (3):
  - University of Virginia Health System, Charlottesville, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Wages NA, Sanders JC, Smith A, Wood S, Anscher MS, Varhegyi N, Krupski TL, Harris TJ, Showalter TN. Hypofractionated Postprostatectomy Radiation Therapy for Prostate Cancer to Reduce Toxicity and Improve Patient Convenience: A Phase 1/2 Trial. Int J Radiat Oncol Biol Phys. 2021 Apr 1;109(5):1254-1262. doi: 10.1016/j.ijrobp.2020.11.009. Epub 2020 Nov 21. PMID 33227441